CLINICAL TRIAL: NCT06717230
Title: Evaluating The Clinical Success And Patient Satisfaction of Digital, Conventional, And Biomimetic Approaches For Restoring Endodontically Treated Teeth: Randomized Controlled Trial.
Brief Title: Digital, Conventional, And Biomimetic Approaches for Restoring Endodontically Treated Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-2024
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital | interventions — EverX Posterior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The child participants and the legal guardian of each participating child and the statistician were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EverX Posterior with Vita Endo-Crowns, EverX Posterior with Bulk-Fill Resin Restorations (Experimental): Biomimetic dentistry leverages modern materials to replicate the biological and mechanical functions of natural teeth, presenting a distinct approach that minimizes the need for extensive tooth reduction and post-placement, particularly advantageous for endodontically treated teeth. Utilizing fiber-reinforced composites, this technique aims to strengthen the dentin-resin bond and evenly distribute occlusal forces across the restoration. By closely adhering to the intact tooth's natural contours and functionality, biomimetic restorations not only preserve more of the natural tooth structure but also reduce stress and strain within the restored tooth. This approach enhances longevity and minimizes the risk of bond failure, with any necessary repairs being straightforward and contributing to the restoration's sustainability.
  Interventions: Other: EverX Posterior
- Lithium Disilicate Endo-Crowns (Active Comparator): conventional restoration for endodontically treated teeth
  Interventions: Other: EverX Posterior

INTERVENTIONS:
Other: EverX Posterior — Restoration

SUMMARY:
Endocrowns are preferred over the post-retained crown, especially at a young age for many reasons; they allow better gingival health and care due to placement of the supragingival margin, have greater fracture resistance limiting the risk for root fracture, thus improving the long-term prognosis of ETMs and has a superior ability to restore ETMs with short crowns, calcified root canals, and thin roots. Furthermore, using CAD/CAM technology facilitates Endocrowns preparation making it simpler with less invasive techniques that can be prepared, fabricated, and cemented in a single visit. The high demand for permanent, esthetic, and conservative restorations has directed clinicians to restore permanent ETMs at a young age with Endo crowns as final coronal restorations.

In addition, Biomimetic dentistry leverages modern materials to replicate the biological and mechanical functions of natural teeth, presenting a distinct approach that minimizes the need for extensive tooth reduction and post-placement, particularly advantageous for endodontically treated teeth. Utilizing fiber-reinforced composites, this technique aims to strengthen the dentin-resin bond and evenly distribute occlusal forces across the restoration. By closely adhering to the intact tooth's natural contours and functionality, biomimetic restorations not only preserve more of the natural tooth structure but also reduce stress and strain within the restored tooth. This approach enhances longevity and minimizes the risk of bond failure, with any necessary repairs being straightforward and contributing to the restoration's sustainability. This study explores the application of fiber-reinforced composites within a biomimetic framework for restoring endodontically treated teeth, aiming to achieve durable and biologically compatible outcomes.

DETAILED DESCRIPTION:
This randomized controlled trial study will evaluate the clinical success of digital, conventional, and biomimetic techniques in restoring endodontically treated mandibular first permanent molars.

Research question:

Are Lithium Disilicate Endo-Crowns, EverX Posterior with Vita Endo-Crowns, and EverX Posterior with Bulk-Fill Resin Restorations Clinically Successful for Restoring Endodontically Treated Mandibular First Permanent Molars?

PICOS:

P: Patients aged ≥15 years with endodontically treated mandibular first permanent molars.

I (1): EverX Posterior with Vita Endo-Crowns I (2): EverX Posterior with Bulk-Fill Resin Restorations C: Lithium Disilicate Endo-Crowns OI: Clinical Success OII: Radiographic Success OIII: Patient satisfaction S: In-Vivo Study

II. Methods

Study Design:

Study Type: Interventional (Controlled Trial) Estimated Enrolment: 42 Teeth Allocation: Randomized Intervention Model: Parallel Assignment Primary Purpose: Treatment Official Title: Evaluating the Clinical Success and Patient Satisfaction of Digital, Conventional, and Biomimetic Approaches For Restoring Endodontically Treated Teeth: Randomized Controlled Trial Estimated Study Start Date: September 2024 Estimated Primary Completion Date: October 2025

Trial design:

The study is a randomized controlled trial (RCT) where 2 arm parallel groups with a 1:1 allocation ratio were compared. The child participants and the legal guardian of each participating child and the statistician were blinded.

Outcome Measures:

1. Primary outcome: Clinical success/ survival [Time Frame: 12 months].

   * Clinical success will be evaluated using (a modified version of the United States Public Health Service (USPHS) criteria which involves the assessment of margins, anatomic form, surface texture, and shade match. (Rate: Alfa, Bravo, Charlie)
   * Each parameter will be assessed using visual and tactile observations (probe, mirror, and dental floss).
   * Treatment will be considered a failure if the restoration had to be remade for any reason including debonding, fracture, or poor appearance, during the 12-month observation period.
2. Secondary outcomes: [Time Frame: 12 months].

   * The radiographic assessment: will involve periapical radiographs to assess the presence of marginal defects, recurrent caries on the same tooth, caries in adjacent teeth, and the presence of periapical infection. (Binary: yes or no)
   * At the checkup visits (3, 6, 9, 12 months), will take standardized photographs, and radiographs, and the restorations will be clinically and radiographically evaluated by an independent and calibrated clinician.
   * Patient-centred outcomes to the restoration: Patient's satisfaction questionnaire. (19) Patient satisfaction in terms of the shape and shade of the end crown, their ability to chew and ﬂoss, and their overall satisfaction with the restoration provided will be assessed on a ﬁve-category visual-analogue scale (extremely satisﬁed, satisﬁed, neutral, dissatisﬁed and extremely dissatisﬁed). All data will be anonymously entered and saved into an Excel sheet in a secured computer only accessible by the principal investigator. [Appendix B] Eligibility Criteria

Ages Eligible for Study: Patients aged ≥15 years. Sexes Eligible for Study: All Accepts Healthy Volunteers: Yes

Criteria

Inclusion Criteria:

1. Endodontically-treated molar tooth with significant loss of tooth structure (both marginal ridges lost) requiring cuspal coverage.
2. Patients aged ≥15 years.
3. Controlled dental disease - no active caries or periodontal diseases
4. Patients will be available to be clinically reviewed up to 1 year

Exclusion Criteria:

1. Patients with poor oral hygiene.
2. Teeth with extensive cracks or fractures.
3. Deep subgingival margins (>0.5mm subgingival).
4. Non-restorable teeth.
5. Non-functional teeth (no opposing dentition).
6. Pocket probing depth > 3mm.
7. Mobility.
8. Patients with bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Endodontically-treated molar tooth with significant loss of tooth structure (both marginal ridges lost) requiring cuspal coverage.
* Patients aged ≥15 years.
* Controlled dental disease - no active caries or periodontal diseases
* Patients will be available to be clinically reviewed up to 1 year

Exclusion Criteria:

* Patients with poor oral hygiene.
* Teeth with extensive cracks or fractures.
* Deep subgingival margins (>0.5mm subgingival).
* Non-restorable teeth.
* Non-functional teeth (no opposing dentition).
* Pocket probing depth > 3mm.
* Mobility.
* Patients with bruxism.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success and survival of restoration | 12 months
  * Clinical success will be evaluated using (a modified version of the United States Public Health Service (USPHS) criteria which involves the assessment of margins, anatomic form, surface texture, and shade match. (Rate: Alfa, Bravo, Charlie)
  * Each parameter will be assessed using visual and tactile observations (probe, mirror, and dental floss).
  * Treatment will be considered a failure if the restoration had to be remade for any reason including debonding, fracture, or poor appearance, during the 12-month observation period.

SECONDARY OUTCOMES:
The radiographic assessment | 12 months
  will involve periapical radiographs to assess the presence of marginal defects, recurrent caries on the same tooth, caries in adjacent teeth, and the presence of periapical infection. (Binary: yes or no)
  • At the checkup visits (3, 6, 9, 12 months), will take standardized photographs, and radiographs, and the restorations will be clinically and radiographically evaluated by an independent and calibrated clinician.
Patient-centred outcomes to the restoration | 12 months
  Patient satisfaction in terms of the shape and shade of the end crown, their ability to chew and ﬂoss, and their overall satisfaction with the restoration provided will be assessed on a ﬁve-category visual-analogue scale (extremely satisﬁed, satisﬁed, neutral, dissatisﬁed and extremely dissatisﬁed).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - MSA University, El-Sheikh Zayed City, Giza Governorate
  - MSA University, Giza

IPD SHARING:
Plan to Share IPD: Undecided